CLINICAL TRIAL: NCT05341063
Title: The Effect of OnlineEducation Given to Individuals With Newly Diagnosed Type 2 Diabetes on Metabolic Control, Self-Care and Health Literacy
Brief Title: New Diagnosed Type 2 Diabetes - Online Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2021/294
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Following the first meeting after the pre-tests, a weekly training was created via Zoom. Diabetes education presentations prepared beforehand were explained in two parts in each training. Training interventions were carried out weekly over Zoom for 4 weeks, lasting approximately 40 minutes. Patients' questions were answered.
  Interventions: Behavioral: Online Education
- Control Group (Experimental): The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Online Education — Diabetes education presentations prepared beforehand were explained in two parts in each training. Training interventions were carried out weekly over Zoom for 4 weeks, lasting approximately 40 minutes. Patients' questions were answered.
  Two months after the training was completed, the current routine analysis results of the participants were taken again, and height and weight measurements were made with the same measurement tools. Participants were allowed to fill in the data collection forms again.
  Arms: Intervention Group
Other: Control Group — The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Arms: Control Group

SUMMARY:
To determine the effect of online education given to individuals with newly diagnosed type 2 diabetes on metabolic control, self-care and health literacy. A randomized controlled trial. This study was conducted with 95 new diagnosed diabetes patients in the Endocrine Polyclinic of a university hospital. Personal Information Form, Diabetes Self-Care Activities Scale and Health Literacy Scale were used to evaluate the data. SPSS 21 program was used in the analysis of the data and a p<0.05 level was considered significant.

DETAILED DESCRIPTION:
Participants were randomized into both groups (intervention and control). The Consolidated Standard of Reporting Trials-CONSORT 2010-guidelines were used to conduct a randomized controlled trial. Sample size was estimated using the G*POWER software tool, based on 80% power and 95% confidence interval. A minimum of 45 individuals in each group were needed to determine the difference in the mean of the measurements (10% more calculated for the probability of sample loss). Between the data collection dates, 248 patients were reached and invited to participate in this study. 78 patients did not meet the inclusion criteria and 70 patients refused to participate. A total of 100 eligible patients were randomized; 50 were assigned to the intervention group and 50 to the control group. After reaching the targeted number, data collection forms were filled in. The participants were then randomly randomized into control and intervention groups in the computer program. Until the randomization was made, it was not known in which groups the individuals were. Randomization was performed after the target number was reached. The first diabetes self-management training was given to all patients by diabetes education nurses face-to-face in the outpatient clinic.

After the study objectives were stated and informed consent was obtained from the study participants, face-to-face interviews by trained interviewers were used to complete the questionnaires. The interviews lasted 20-25 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Type 2 diabetes mellitus for at most one year
* Be between the ages of 18-65
* Being on oral antidiabetic and/or insulin therapy
* Have a smart phone
* Volunteer to participate in the study
* Hearing that interferes with communication
* Sensory loss such as speech
* Psychiatric problem

Exclusion Criteria:

* Illiterate
* Have a physical, cognitive or mental disability to answer questions
* Individuals with type 2 DM who did not volunteer to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The Diabetes Self-Care Activities Questionnaire | 5 minute
  The Diabetes Self-Care Activities Questionnaire was developed by Toobert and Glasgow to determine the self-care activities of individuals with diabetes. The Turkish validity and reliability of the questionnaire were conducted by Kav et al. (2010) and the total Cronbach alpha value was found 0.72. The tool contains 11 items, which measure the frequency of performing dia- betes self-care activities over the last seven days including diet, exercise, blood glucose testing, foot care and tobacco use. The scale total score ranges between 0-7. Higher scores indicate more self-care activities.
Health Literacy Scale | 5 minute
  It is a 4-point Likert type scale consisting of 14 items and three parts, developed by Ishikawa et al. (2008). The scale was developed to measure the functional, interactive and critical health literacy of individuals with chronic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Aydemir, Dr, Study Chair — Akdeniz University Hospital
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Agarwal P, Mukerji G, Desveaux L, Ivers NM, Bhattacharyya O, Hensel JM, Shaw J, Bouck Z, Jamieson T, Onabajo N, Cooper M, Marani H, Jeffs L, Bhatia RS. Mobile App for Improved Self-Management of Type 2 Diabetes: Multicenter Pragmatic Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 10;7(1):e10321. doi: 10.2196/10321. PMID 30632972
- [Result] Park J, Kim SH, Kim JG. Effects of message framing and health literacy on intention to perform diabetes self-care: A randomized controlled trial. Diabetes Res Clin Pract. 2020 Mar;161:108043. doi: 10.1016/j.diabres.2020.108043. Epub 2020 Jan 30. PMID 32006642